CLINICAL TRIAL: NCT05786261
Title: Exercise and Plasticity in PD: Functional and Structural Evidence in the Cortex and the Spinal Cord
Brief Title: Exercise and Plasticity in Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PD180091
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group MIRT (Experimental): Task 1a: Assessing the effect of MIRT on cortical plasticity tested with rPAS Task 1b: Assessing the effect of MIRT on structural cortical plasticity and brain connectivity tested with MRI Task 1c: Assessing the effect of MIRT on movement-related beta modulation Task 1d: Assessing the effects of MIRT on motor skills formation with reaching tasks Task 1e: Assessing the effects of MIRT on EEG correlates of motor skills formation Task 2a: Assessing the effect of MIRT on muscle synergies during gait Task 2b: Assessing the effect of MIRT on muscle synergies during reaching movements Task 3a: Assessing the effect of MIRT on sleep microstructure
  Interventions: Device: experimental group MIRT; Device: EEG task rTMS, fMRI
- control group (Active Comparator): EEG con task, Gait Analysis, fMRI, rTMS,
  Interventions: Device: EEG task rTMS, fMRI

INTERVENTIONS:
Device: experimental group MIRT — Task 1a: Assessing the effect of MIRT on cortical plasticity tested with rPAS Task 1b: Assessing the effect of MIRT on structural cortical plasticity and brain connectivity tested with MRI Task 1c: Assessing the effect of MIRT on movement-related beta modulation Task 1d: Assessing the effects of MIRT on motor skills formation with reaching tasks Task 1e: Assessing the effects of MIRT on EEG correlates of motor skills formation Task 2a: Assessing the effect of MIRT on muscle synergies during gait Task 2b: Assessing the effect of MIRT on muscle synergies during reaching movements Task 3a: Assessing the effect of MIRT on sleep microstructure
  Arms: experimental group MIRT
Device: EEG task rTMS, fMRI — EEG task rTMS, fMRI

SUMMARY:
We will study the effects of intensive rehabilitation in PD on plasticity with a multimodal approach. We will define first, whether exercise in PD restores the potentiation of the motor cortex to normal levels with both 5 Hz-rTMS PAS and beta modulation and whether such improvements are accompanied by structural changes studied with diffusion MRI tractography and network analysis (Aim 1). With the study of muscle synergies and spatiotemporal organization of the spinal motoneuronal output during gait and reaching movements we will define the presence of functional changes in spinal cord mechanisms and connectivity and whether such changes are global or involve selective districts (Aim 2). Finally, we will study post-exercise changes in sleep pattern, as sleep is impaired in PD and plays a crucial role in the definition of plasticity-related phenomena (Aim 3). This project will generate breakthrough data on the mechanisms of exercise, novel biomarkers to monitor efficacy of treatments and thus, possibly leading to better restorative, disease-modifying and symptomatic therapies for PD.

DETAILED DESCRIPTION:
We will study the effects of intensive rehabilitation in PD on plasticity with a multimodal approach. We will define first, whether exercise in PD restores the potentiation of the motor cortex to normal levels with both 5 Hz-rTMS PAS and beta modulation and whether such improvements are accompanied by structural changes studied with diffusion MRI tractography and network analysis (Aim 1). With the study of muscle synergies and spatiotemporal organization of the spinal motoneuronal output during gait and reaching movements we will define the presence of functional changes in spinal cord mechanisms and connectivity and whether such changes are global or involve selective districts (Aim 2). Finally, we will study post-exercise changes in sleep pattern, as sleep is impaired in PD and plays a crucial role in the definition of plasticity-related phenomena (Aim 3)

ELIGIBILITY:
Inclusion Criteria:

Idiophatic Parkinson Disease

* H&Y stage I-II stable medication

Exclusion Criteria:

* Severe comorbid medical illness (diabetes, heart disease, hypertension); history of known causative factors (encephalitis or neuroleptic treatment); other neurologic disability; chronic treatment for sleep complaints; history of seizure, including febrile seizures, family history of epilepsy; pacemakers, neurostimulators, tattoos, metal foreign bodies in the head area; recurrent visual hallucinations; fluctuating cognition, attention or alertness; depression (HAMD> 12) or dementia (MMSE <24).

Controls will be age- and education- matched subjects.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
functional magnetic resonance | 1 month
  assessment of the functional and structural plasticity changes after MIRT

SECONDARY OUTCOMES:
EMG | 1 month
  muscle synergies and spatiotemporal organization of the spinal motoneuronal output during gait and reaching movements we will define the presence of functional changes in spinal cord mechanisms and connectivity and whether such changes are global or involve selective districts

OTHER OUTCOMES:
PS EEG | 1 month
  we will study post-exercise changes in sleep pattern, as sleep is impaired in PD and plays a crucial role in the definition of plasticity-related phenomena

CONTACTS AND LOCATIONS:
Overall Officials: felice ghilardi, MD, Principal Investigator — City College of New York, New York, NY
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: No
Principal Investigator